CLINICAL TRIAL: NCT05003687
Title: Interventional, Randomized, Double-Blind, Sequential-Group, Placebo-Controlled, Single-Ascending Oral Dose Study Investigating the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Properties of Lu AG06474 and Open-Label, Cross-Over Study to Investigate Intra-Subject Variability and the Effect of Food in Healthy Young Men
Brief Title: Safety and Tolerability of Lu AG06474 in Healthy Young Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 19702A
Record Dates: First submitted 2021-08-06; First posted 2021-08-12 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Part A: randomized, double-blind, sequential. Part B: randomized, open-label, cross-over.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Single Dose of Lu AG06474 or Placebo (Experimental): Participants will receive single oral dose of Lu AG06474 or placebo.
  Interventions: Drug: Lu AG06474; Drug: Placebo
- Part B: Repeated Dose of Lu AG06474 and Food Interaction (Experimental): Participants will receive a single oral dose of Lu AG06474 in each dosing period (Period 1, 2, and 3) in the following sequence:
  Sequence B1: Fed - Fasting- Fasting
  Sequence B2: Fasting- Fed - Fasting
  Sequence B3: Fasting- Fasting - Fed
  Interventions: Drug: Lu AG06474

INTERVENTIONS:
Drug: Lu AG06474 — solution, orally (Parts A and B)
Drug: Placebo — solution, orally (Part A only)
  Arms: Part A: Single Dose of Lu AG06474 or Placebo

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of Lu AG06474 and what the body does to Lu AG06474 after swallowing single doses of the drug.

DETAILED DESCRIPTION:
Part A: randomized, double-blind, sequential. Part B: randomized, open-label, cross-over.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a body mass index (BMI) ≥18.5 and ≤30 kilograms (kg)/square meter (m^2) at the Screening Visit and at the Safety Baseline/Baseline Visit.
* The participant is, in the opinion of the investigator, generally healthy based on medical history, a physical examination, vital signs, a safety ECG, and the results of the clinical chemistry, haematology, urinalysis, serology, and other laboratory tests.

Exclusion Criteria:

* The participant has taken disallowed medication <1 week prior to the first dose of study drug or <5 half-lives prior to the Screening Visit for any medication taken.
* The participant has orthostatic hypotension, defined as a decrease in systolic blood pressure ≥20 millimeters of mercury (mmHg) and/or a decrease in diastolic blood pressure ≥10 mmHg from supine to standing, at the Screening Visit or at the Safety Baseline/Baseline Visit.
* The participant has a QTcF interval >450 milliseconds (ms) at the Screening Visit or at the Safety Baseline/Baseline Visit, as calculated by the ECG equipment and evaluated by the investigator.
* The participant has taken any investigational medicinal product <3 months prior to the first dose of study drug.
* The participant has received an injection of COVID-19 vaccination less than 30 days prior to the first dose of study drug.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Parts A and B: Number of participants With Treatment-Emergent Adverse Events | From Baseline to Day 8
Part A: Electrocardiogram (ECG) Parameter (Delta QTcF) at 24 Hours on Day 1 | Day 1
Part A: Change From Pre-Dose Baseline in ECG Parameter (Delta QTcF) at 24 Hours on Day 1 | Pre-dose Baseline (Day -1), Day 1
Part A: Bond-Lader VAS Dimension Scores at Day 4 | Day 4
Part A: Change From Pre-Dose Baseline in the Bond-Lader VAS Dimension Scores at Day 4 | Pre-dose Baseline (Day -1), Day 4
Part A: Percentage of Peripheral Blood Mononuclear Cells (PBMC)-Mediated Hydrolysis of 2-arachidonolylglycerol (2-AG) Ex Vivo (% of Pre-Dose Measurement of Arachidonic Acid [AA]) | From pre-dose to Day 4
Parts A and B: AUC0-inf of Lu AG06474 | From pre-dose to Day 4
  Area under the Lu AG06474 concentration-time curve from time zero to infinity (AUC0-inf)
Parts A and B: Cmax of Lu AG06474 | From pre-dose to Day 4
  Maximum observed plasma concentration for Lu AG06474
Parts A and B: Tmax of Lu AG06474 | From pre-dose to Day 4
  Nominal time corresponding to the occurrence of Cmax of Lu AG06474
Part A: t1/2 of Lu AG06474 | From pre-dose to Day 4
  Apparent elimination half-life of Lu AG06474

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — H. Lundbeck A/S
Locations (1):
- Quotient Sciences Miami, Miami, Florida, United States